CLINICAL TRIAL: NCT05764226
Title: A Clinical Study of Freshly Manufactured 35kDa Hyaluronan Fragment HA35 for Treatment of Chronic Wounds
Brief Title: Freshly Manufactured 35kDa Hyaluronan Fragment HA35 for the Treatment of Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhia Impex LLC (Industry)
Collaborators: Mongolian National University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hui19970909
Record Dates: First submitted 2023-02-16; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Chronic Wounds
Keywords: Hyaluronidase; 35kDa hyaluronan fragment; HA35; Tissue permeability; Chronic wound; Wound healing

STUDY DESIGN:
Intervention Model Description: An open label single arm before and after treatment comparison clinical study
Masking Description: An off-label use of an open label single arm before and after treatment comparison clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35 kDa HA fragment HA35 injection (Experimental): 100 mg of the freshly made 35 kDa low molecular weight hyaluronan fragment HA35 was injected into the tissue under the heath skin immediately surrounding the chronic wounds
  Interventions: Drug: HA35(L20200708MP07707, Ministry of Health, Mongolia)was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089)

INTERVENTIONS:
Drug: HA35(L20200708MP07707, Ministry of Health, Mongolia)was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089) — One hundred milligrams of the freshly made 35 kDa low molecular weight HA fragment HA35 was injected into the tissue under the heath skin immediately surrounding the chronic wounds once a day for 10 days.
  Other Names: HA35

SUMMARY:
In this research, the patients with chronic wounds accompanied by pain were treated by injecting freshly manufactured tissue permeable hyaluronan fragment HA35 into the tissue under the heath skin immediately surrounding the chronic wounds.

DETAILED DESCRIPTION:
Chronic wounds are wounds or ulcers that do not heal properly and are generally classified as venous, arterial, diabetic, traumatic, and pressure chronic wound. Persistent chronic inflammation is a hallmark for chronic wound or trauma and is also often associated with inflammatory and neuropathic pain.

Injections of high molecular weight hyaluronan HA into joint cavity have been used for many years in treatment of joint pain as well as associated inflammation. Still, due to the high viscosity and poor tissue permeability of high molecular weight HA, it is unsuitable for treating chronic wound or trauma pain and the associated inflammation. In this study, the investigators found that hyaluronidase PH20 could cleave high molecular weight hyaluronan into 35kDa low molecular weight hyaluronan fragment HA35. The freshly-made hyaluronan fragment HA35 had great tissue permeability compared with high molecular HA. Our previous clinical studies (http://www.clinicaltrials.gov) have shown freshly-made hyaluronan fragment HA35 effectively treating shoulder, neck and back pain as well as the severe pain associated with shingles. In this study, the tissue-permeable 35kDa hyaluronan fragment HA35 was freshly manufactured by mixing hyaluronidase PH20 injectable solution and high-molecular-weight hyaluronan HA injectable solution. The therapeutic effect of the tissue-permeable hyaluronan fragment HA35 for treatment of pain associated chronic wounds was studied in a single-arm off-label used, before and after treatment comparison, clinical study similar to others.

Both recombinant human hyaluronidase PH20 (Hylenex, Halozyme Inc) and bovine testis-derived hyaluronidase PH20 (H31022111) are able to cleave high molecule weight hyaluronan into 35 kDa hyaluronan fragments HA35 (L20200708MP07707, Ministry of Health, Mongolia). This clinical study uses 35kDa low molecular weight hyaluronan fragment HA35 which was freshly manufactured by mixing bovine testis-derived hyaluronidase PH20 injection (H31022111) with high molecular weight hyaluronan HA injection (H20174089) for 20 minutesat at room temperature.

In this study, 20 hospitalized patients with chronic wounds accompanied by pain were treated with the freshly manufactured 35 kDa low molecular weight hyaluronan fragment HA35. There were 8 patients with diabetic chronic wounds, 4 patients with chronic venous wounds, 2 patients with chronic arterial wounds, 6 patients with traumatic and chronic pressure wounds. Among these patients, there are 12 males and 8 females, having average age of 55±10 years. The creteria for the chronic wound in this study were the wound that has not been healed more than 3 months. All the chronic wounds were associated with significantly pain. All the wounds were clinically presented by surface darkenes and purulent secretions on the wounds, and darkness, redness, swelling and dryness and broken surface of the skin surrounding the wounds. This study is an open-label clinical study in which no information is withheld from participantes and investigators. In this study, the therapeutic effect was studied by comparison of those of before and after treatment in a single-arm study. The pain associated with the wounds and degree of healing of the wounds including the size of fresh granulation area on the wound, the degree of darkness or redness, dryness and broken surface of the skin surrounding the wound, and the size of the wound were observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. The chronic wounds of painful diabetic wounds, venous wounds, arterial wounds, traumatic and pressure wounds which had not been closed more than 3 months.
2. All the chronic wounds were clinically presented by surface darkeness and purulent secretions on the wounds, and darkness or redness, swelling, dryness and broken.
3. Surface of the skin immediately surrounding the wounds.
4. Subject agrees to be compliant with study related visit and treatment schedule.
5. Written informed consent.

Exclusion Criteria:

1. History of wound healing abnormalities or a medical condition that is known to be associated with abnormal wound healing.
2. Subjects with any known coagulation disorder.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
The pain score | 24 hours
  Primary outcome in this clinical study is the pain score of all kinds of chronic wound, inclouding diabetic chronic wounds, chronic venous wounds, chronic arterial wounds ,traumatic and chronic pressure wounds. The pain scale is a tool typically employed by clinicians for pain assessment. Participants use a specially designed scale to do self-assessment for pain intensity. Each participant rates the pain on a scale of 0-10 where 0 represents "no pain" while 10 represents "the most intensive pain". In this study, the pain intensity was assessed before and after the treatment.

SECONDARY OUTCOMES:
The self-quantitative assessment scale | 10 days
  The secondary outcome measure is the self-quantitative assessment scale of chronic trauma signs which is a modified version of the Pain Scale. The chronic trauma signs include darkness or redness, dryness and broken skin surface, fresh granulation growth area of the wounds, and the size of the wounds.
  The participant rates the intensity level using scale of 0-10 where 0 represents "no dryness and broken surface" while 10 represents "the most intensive dryness and broken surface".
  The participant rates the intensity level using scale of 0-10 where 0 represents "no fresh granulation growth" while 10 represents "the most intensive fresh granulation growth" which equals 100% of wound surface area covered by the fresh granulation growth.
  The participant rates the size or area using scale of 0-10 where 0 represents "no wound size change at all" while 10 represents wound 100% closed or healed".

CONTACTS AND LOCATIONS:
Locations (1):
- Far East Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: published precinical study and international granted patent
Access Criteria: Anti-Inflammatory Effects of the 35kDa Hyaluronic Acid Fragment (B-HA/ HA35); APPLICATION OF LOW-MOLECULAR-WEIGHT HYALURONIC ACID(LMW-HA) FRAGMENTS(INJECTION) WO/2017/186088 US20200254005 EP3479830 AU2017255833 CA3049286
URL: http://www.dovepress.com/articles.php?article_id=80993；https://patentscope.wipo.int/search/en/detail.jsf?docId=CA249072967&_cid=P22-LDWT33-38680-1

REFERENCES:
- [Result] Jia X, Shi M, Wang Q, Hui J, Shofaro JH, Erkhembayar R, Hui M, Gao C, Gantumur MA. Anti-Inflammatory Effects of the 35kDa Hyaluronic Acid Fragment (B-HA/HA35). J Inflamm Res. 2023 Jan 13;16:209-224. doi: 10.2147/JIR.S393495. eCollection 2023. PMID 36686276
- [Result] APPLICATION OF LOW-MOLECULAR-WEIGHT HYALURONIC ACID(LMW-HA) FRAGMENTS(INJECTION) WO/2017/186088 US20200254005 EP3479830 AU2017255833 CA3049286
- See also: Related Info — http://patentscope.wipo.int/search/en/detail.jsf?docId=CA249072967&_cid=P22-LDWT33-38680-1